CLINICAL TRIAL: NCT06635772
Title: A Randomized, Multicenter, Open-label, Active-control Study of the Efficacy and Safety of HS-10390 for the Treatment of Immunoglobulin a Nephropathy
Brief Title: A Study of the Effect and Safety of HS-10390 in the Treatment of Patients with Primary IgA Nephropathy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-10390-201
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Immunoglobulin a Nephropathy
Keywords: Immunoglobulin A Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Irbesartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HS-10390; high dose (Experimental): HS-10390; high dose
  Interventions: Drug: HS-10390
- HS-10390; low dose (Experimental): HS-10390; low dose
  Interventions: Drug: HS-10390
- irbesartan (Active Comparator): Irbesartan will be administered daily as a 150-mg oral tablet. For patients who tolerate the initial dose of 150 mg after 2 weeks will increase their dose to 300 mg
  Interventions: Drug: Irbesartan

INTERVENTIONS:
Drug: HS-10390 — HS-10390 will be administered daily
  Arms: HS-10390; high dose; HS-10390; low dose
Drug: Irbesartan — Irbesartan will be administered daily as a 150-mg oral tablet. For patients who tolerate the initial dose of 150 mg after 2 weeks will increase their dose to 300 mg
  Arms: irbesartan

SUMMARY:
This study will evaluate the efficacy and safety of HS-10390 in subjects with primary IgA nephropathy, and explore the optimal dose for the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 18 and 65 years age.
* Biopsy-proven primary IgA nephropathy.
* Currently on stable dose of ACEI and/or ARB therapy, for at least 12 weeks prior to screening (the patient's maximum tolerated dose and is at least one-half of the maximum labeled dose).
* Average 24-hour urine total protein ≥ 0.75 g/24 h at screening.
* Estimated GFR (using the CKD-EPI 2009) ≥ 30 mL/min per 1.73 m^2 at screening.
* Systolic BP between 100 and 150 mmHg and diastolic BP between 60 and 100 mmHg.

Exclusion Criteria:

* IgA nephropathy secondary to another condition
* IgA nephropathy with rapid decline of renal function; Kidney pathology indicated that more than 50% of the glomerulus had large crescent body formation, which may affect the study results; Tubule atrophy - interstitial fibrosis of more than 50%;
* Chronic kidney disease (CKD) in addition to IgAN
* Patients treated with any systemic non-biologic immunosuppressive drugs (including systemic corticosteroids) within 12 weeks prior to randomizing；
* Require any prohibited medications prior to randomizing;
* Exposure to an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to screening
* History of organ transplantation, with exception of corneal transplants
* Platelet< 100×109/L or hemoglobin value < 90 g/L) or Hematocrit value < 27% (0.27 V/V) at Screening
* Elevations of transaminases (ALT and/or AST) >2 times upper limit of normal or total bilirubin and/or direct bilirubin exceeding 1.5 times the upper limit of normal (ULN) at screening
* Potassium >5.5 mmol/L at Screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 24-hour urine protein at Week 12 | up to week 12
  The change in urine protein: creatinine ratio (UPCR) from baseline to Week 12

SECONDARY OUTCOMES:
Change from baseline in 24-hour urine protein (UPCR) | up to Week 12
  The change in urine protein: creatinine ratio (UPCR) from baseline
Change from baseline in 24-hour urine protein(UACR) | up to Week 12
  The change in urine albumin: creatinine ratio (UACR) from baseline
Change from baseline in 24-hour urine protein | up to Week 12
  The change in urine protein excretion from baseline
Proportion Change from baseline in 24-hour urine protein | up to Week 12
  The proportion of patients with urinary protein equivalent of < 0.3 g/24 hours
change from baseline in Estimated Glomerular Filtration Rate | up to Week 12
  change from baseline in Estimated Glomerular Filtration Rate (eGFR)
Number of subjects with adverse events (AEs) | up to Week 12
  Type, incidence, severity, seriousness, and relatedness of AEs will be collected
Plasma Concentration of HS-10390 | up to Week 12
  Blood samples will be collected for the measurement of plasma concentrations of HS-10390

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China